CLINICAL TRIAL: NCT06194435
Title: Impact of Teleexercise and Remote Assessments in Rotator Cuff Syndrome: A Comparative Trial
Brief Title: Teleexercise for Rotator Cuff Syndrome: A Comparison
Acronym: TFRCSAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Selkin Yılmaz Muluk, MD, Physical Therapy and Rehabilitation specialist, Antalya Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Antalya Ataturk State Hospital
Record Dates: First submitted 2023-11-30; First posted 2024-01-08 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Rotator Cuff Syndrome
Keywords: rotator cuff syndrome; telemedicine; teleexercise; asynchronous video
MeSH Terms: interventions — Health

STUDY DESIGN:
Intervention Model Description: Study Design: This study utilizes a randomized controlled parallel-design approach to evaluate the effectiveness of telemedicine methods in treating RCS compared to traditional in-person methods.
  Participants: The study will include 76 participants aged 40 to 60 years diagnosed with RCS, confirmed through shoulder MRI, and unresponsive to conservative treatments. They are randomly assigned to two groups.
  Intervention Group/Telemedicine Group: Remote assessments, video exercise program, and virtual follow-ups.
  Control Group: In-person assessments, exercise program, and follow-ups.
  Data Collection: Comprehensive documentation of clinical diagnoses and demographics, informed consent, and outcome measures (Quick-DASH and Numeric-VAS) are collected.
  Outcome Measures: The study assesses pain levels, functional recovery, and overall treatment outcomes.
  Analysis: Statistical analysis is conducted to compare treatment effectiveness between the two groups.
Who Masked: Outcomes Assessor
Masking Description: The person conducting the statistical analysis will be unaware of group identities, she will perform the data analysis without knowledge of which group received which treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Group: Remote Assessments and Asynchronous Exercise Guidance (Experimental): For the Telemedicine Group, the study initiates with a video call from the physician on day one via FaceTime or WhatsApp. During these calls, patients will receive guidance and complete Quick-DASH questionnaire and numeric-VAS scale. On the same day, they will also receive an exercise video and an exercise diary via WhatsApp. Follow-up video calls on the 7th day will serve as reminders and allow patients to ask questions. The final video call, scheduled for the 15th day, will involve completing the same questionnaire and scale. After this last remote interaction, patients will send photos of their completed exercise logs to the physician via WhatsApp for adherence tracking.
  Interventions: Other: Remote Monitoring of Participant Progress and Well-being via Video Calls
- Control Group: In-Person Assessments in Clinic and Exercise Brochure (Active Comparator): For the Control Group, the study begins with an in-person visit to the physician on day one. During this visit, patients will receive guidance, complete Quick-DASH questionnaire and numeric-VAS scale, and be provided with an exercise brochure. Additionally, patients will receive an exercise diary on the same day to record their exercise sessions. Follow-up visits to the physician's office at the hospital on the 7th day will serve as reminders and opportunities for patients to ask questions. On the 15th day, patients will revisit the hospital to complete the same questionnaire and scale. We will also assess the time spent and economic burden associated with hospital visits. Furthermore, exercise diaries will be collected for adherence tracking and progress evaluation.
  Interventions: Other: Face-to-Face Clinic-based Monitoring of Participant Progress and Well-being

INTERVENTIONS:
Other: Remote Monitoring of Participant Progress and Well-being via Video Calls — Participants with Rotator Cuff Syndrome undergo remote evaluations via video calls with a physician. On the same day, they receive an asynchronous exercise brochure containing instructions for performing home exercises three times a day. They are also provided with an exercise diary to track their daily exercise sessions. Follow-up assessments and discussions about their condition take place remotely on video calls with the physician on the 7th and 15th days. During the final video call on the 15th day, participants are asked to submit their exercise diaries via WhatsApp for assessment of exercise adherence.
  Other Names: Delivery of Asynchronous Home Exercise Video Through WhatsApp; Monitoring Exercise Adherence Using Exercise Diaries; Evaluating Shoulder Function and Pain Using Questionnaire and Pain Scale After Home Exercise Program
  Arms: Telemedicine Group: Remote Assessments and Asynchronous Exercise Guidance
Other: Face-to-Face Clinic-based Monitoring of Participant Progress and Well-being — Participants with Rotator Cuff Syndrome undergo in-clinic evaluations by a physician, during which they receive an exercise brochure with instructions for performing home exercises three times a day. They are also given an exercise diary to track their daily exercise sessions. On the 7th and 15th days, participants return for follow-up assessments and discussions about their condition. During the final clinic visit, participants are requested to submit their exercise diaries for assessment of exercise adherence.
  Other Names: Hand-Delivery of Home Exercise Brochure; Monitoring Exercise Adherence Using Exercise Diaries; Evaluating Shoulder Function and Pain Using Questionnaire and Pain Scale After Home Exercise Program
  Arms: Control Group: In-Person Assessments in Clinic and Exercise Brochure

SUMMARY:
Rotator Cuff Syndrome (RCS) often lead to shoulder pain and reduced function, creating a demand for alternative treatments. This study examines the effectiveness of remote assessments and tele-exercise compared to traditional in-person methods for treating these injuries. The telemedicine group will receive remote consultations and asynchronous exercise videos, while the control group will have face-to-face meetings and comprehensive information. Follow-up assessments will track exercise compliance for both groups. Additionally, a questionnaire will assess functionality, and pain levels will be evaluated using a pain scale, providing a comprehensive evaluation of treatment outcomes.

DETAILED DESCRIPTION:
This study employs a randomized controlled clinical trial with a parallel design conducted at a hospital-based Physical Therapy and Rehabilitation Clinic. The study is planned to involve 76 voluntary participants.

Inclusion criteria for participants encompass the following: participants must be within the age range of 30 to 65, diagnosed with conditions such as rotator cuff tendinosis, tendinitis, impingement, or partial rupture, confirmed through shoulder MR imaging, have not experienced improvement through conservative methods (e.g., activity restriction, ice application, and analgesics), and must have been referred for physical therapy sessions.

Participants will be randomly assigned to two groups, with efforts to maintain balance in terms of age and gender distribution. Data collection methods include detailed documentation of participants' clinical diagnoses and demographic information (e.g., age, gender, education level, occupation, dominance of the affected side, and whether the occupation involves physical labor or heavy lifting).

Before the study commences, all participants will receive comprehensive explanations of the study's objectives, provide informed consent by signing consent forms, and share their contact information for communication purposes. Participants will be informed of their rights to discontinue treatment at any point and to reach out to the researcher with questions or concerns during the study.

Participants in the Exercise Group will have face-to-face assessments at the clinic on the first day. This includes completing the Quick- Disabilities of the Arm, Shoulder and Hand (Quick- DASH) questionnaire and the Numeric Visual Analog Scale (VAS) for pain assessment. They will receive information about their condition, a brochure containing a home exercise program, and an exercise diary to record exercise details. Follow-up assessments will occur on the 7th and 15th days at the clinic.

Participants in the Telemedicine Group will have a different approach. On the first day of the study, they will have video calls through FaceTime or WhatsApp. The Quick-DASH questionnaire and Numeric VAS scale will be administered and they will receive information about their condition. Subsequently, a pre-recorded video comprising the home exercise program, along with an exercise diary to record exercise details, will be sent to them via WhatsApp. Follow-up assessments will occur on the 7th and 15th days through video calls. Both groups will receive regular follow-up phone calls to collect their VAS scores at the 6th-month mark.

The Quick-DASH questionnaire assesses upper extremity function, including functionality, pain, symptoms, and quality of life. It consists of 11 questions, each scored on a scale. The Numeric VAS pain scale measures pain intensity on a scale of 0 to 10.

The exercise brochure includes exercise descriptions and visual demonstrations aimed at improving joint range of motion, adapted from programs provided by the American Academy of Orthopaedic Surgeons.

The exercise diary provided to participants consists of a table with three columns for each day, spanning 15 days in total. Each day is divided into three time slots: morning, noon, and evening. Participants will be instructed to mark the relevant box when they complete the exercises at the specified times, and if they do not perform the exercises during that particular time slot on a given day, they should leave the box empty.

This methodology aims to assess the impact of telemedicine methods on the treatment outcomes of RCS patients compared to traditional methods, as well as to improve patients' access to treatment and enhance the efficiency of healthcare resources.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of rotator cuff tendinosis, tendinitis, impingement, or partial muscle rupture confirmed by shoulder MRI,
* Not benefiting from conservative methods such as activity restriction, ice application and analgesics, being referred to physical therapy sessions,
* Having single-sided shoulder problem, possessing the ability to understand and perform prescribed exercises,
* Having the cognitive and psychological capacity to read and interpret brochures, being familiar to smartphones for accessing digital exercise materials,
* Having internet access.

Exclusion Criteria:

* Cognitive impairment,
* Bilateral rotator cuff syndrome,
* Total rupture of rotator cuff muscle,
* Previous fractures or surgeries on the same shoulder,
* Shoulder instability,
* Visual impairments,
* Extremity amputations,
* Advanced cancer and complicated diabetes,
* Recent injections to the same shoulder within the last 6 months,
* Having received physical therapy or home exercise advice within the last 6 months,
* Lacking personal smartphones or internet access,
* Undergoing cancer treatment.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Pain Levels | At the first day, the 15th day and the 6th month of the study.
  Assessments of pain intensity using the numeric-Visual Analog Scale (VAS). The numeric-VAS typically ranges from 0 to 10, with 0 representing no pain or symptom and 10 representing the worst imaginable pain or symptom. The highest score on the VAS is 10, indicating the most severe pain or symptom.
Functional Recovery | At the first day and the 15th day of the study.
  Evaluation of upper extremity function using the Quick-Disabilities of Arm, Shoulder, Hand (DASH) questionnaire. The Quick-DASH score can range from 0 to 100, with higher scores indicating more severe disability or symptoms. A score of 0 would mean no disability or symptoms, while a score of 100 would suggest the most severe disability or symptoms. Generally, a lower Quick-DASH score represents better functioning and less disability.
Exercise Adherence | From the first day till the 15th day of the study (15 days time frame).
  Monitoring and recording participants' adherence to the prescribed home exercise program through exercise diaries. This would involve tracking the frequency and consistency of exercise performance.

SECONDARY OUTCOMES:
Patient Satisfaction with Likert Satisfaction Scale | From the first day till the 15th date of the study (15 days time frame).
  Gathering feedback from participants on their satisfaction with the assigned treatment approach for shoulder pain using a Likert scale of satisfaction, where they rate their satisfaction level from 1 (Very Dissatisfied) to 5 (Very Satisfied).
Evaluating Travel Distance and Time for Control Group In-Person Hospital Visits | Data will be collected on the first day of the study.
  Assessing Travel Distance and Time for Control Group Hospital Visits: Participants will provide details of their single-day round-trip travel from home to the hospital and back, including kilometers traveled and minutes spent. This data will be used to calculate the economic burden and time commitment associated with in-person hospital visits.

CONTACTS AND LOCATIONS:
Overall Officials: Selkin Yılmaz, Principal Investigator — Antalya Ataturk Devlet Hastanesi
Locations (1):
- Selkin Yılmaz Muluk, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Our plan is to share individual participant data collected during this study with qualified researchers and institutions for the purpose of promoting transparency and furthering scientific research.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 months after study completion
Access Criteria: Access to the individual participant data will be granted to qualified researchers, institutions, or individuals who submit a formal request.

REFERENCES:
- [Background] Harms S, Kobusingye O. Factors that influence the use of rehabilitation services in an urban Ugandan hospital. Int J Rehabil Res. 2003 Mar;26(1):73-7. doi: 10.1097/00004356-200303000-00012. PMID 12601273
- [Background] Amorese AJ, Ryan AS. Home-Based Tele-Exercise in Musculoskeletal Conditions and Chronic Disease: A Literature Review. Front Rehabil Sci. 2022 Feb 24;3:811465. doi: 10.3389/fresc.2022.811465. eCollection 2022. PMID 36188988
- See also: 'Rotator Cuff and Shoulder Conditioning Program' of American Academy of Orthopaedic Surgeons. — https://orthoinfo.aaos.org/globalassets/pdfs/2017-rehab_shoulder.pdf